CLINICAL TRIAL: NCT05835531
Title: Evaluation of the Efficacy and Safety of Midline Venous Catheters
Acronym: MVC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital El Cruce (Other)
Responsible Party: Principal Investigator, Nestor Pistillo, UTIA, Hospital El Cruce
Other Study IDs: 026/2022
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Midline Catheter
Keywords: infusion therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Catheters comparation — Assessment of incidence of complications associated with midline catheters
  Other Names: MIDLINE VENOUS CATHETERS

SUMMARY:
Central venous catheters are fundamental tools in medical practice, but their use carries frequent local and systemic complications, with bloodstream infection (bacteremia) and thrombus formation being the most frequent and serious. Both complications prolong hospitalization time, increase morbidity, mortality, and hospital costs. Medium access peripheral venous catheters (MC) are a low-cost, easy-to-place, and highly-durable option that offers greater patient comfort and less pain, among other advantages. The objective of this study is to determine if the implementation of a team specialized in the placement of midline (CM) catheters reduces the incidence of infections associated with central venous catheters, decreases the cost of hospitalization, and preserves venous capital in patients admitted to ICU.

DETAILED DESCRIPTION:
Central venous catheters are fundamental tools in medical practice, but their use carries frequent local and systemic complications, with bloodstream infection (bacteremia) and thrombus formation being the most frequent and serious. Both complications prolong hospitalization time, increase morbidity, mortality, and hospital costs. Promoting policies to prevent catheter-associated infections (CAIs) not only reduces the number of complications but is also essential to mitigate and control the development of multidrug-resistant organisms. The mechanism by which catheters become colonized is multifactorial and complex. Mainly, bacteria access the catheter through three access routes: 1) migration of superficial organisms that follow the path of the catheter until they colonize its tip. Generally, this extraluminal form of colonization causes bacteremia in the first days of catheterization. 2) The intraluminal route is the most frequent form of colonization. Inadequate cleaning of system connections, especially in multiple-lumen and multiple-path catheters, allows bacteria to enter after the first week of use. The third colonization route is rare and is due to hematogenous seeding of bacteria from a distant focus of infection or intrinsic contamination of the infused fluid. Other factors that also favor catheter colonization are the type of material (Teflon is less friendly to the vein), the number of lumens (directly proportional to the risk of infection), the nutritional and immunological deterioration of the individual, the type of infusion administered and the insertion site.

Medium access peripheral venous catheters (MC) are a low-cost, easy-to-place, and highly-durable option that offers greater patient comfort and less pain, among other advantages. They are placed using the Seldinger surgical technique at the foot of the bed, in a simple manner, and under ultrasound guidance. The catheter enters through a peripheral vein near the elbow crease and its tip is positioned at the level of the axillary vein, facilitating the infusion of drugs with an osmolarity <600 mOsm, pH range of 5 to 9, and blood derivatives. The success rate of the procedure is almost 100%, particularly if an expert performs the catheterization.

Midline catheters are an intermediate type of catheter between peripheral and central lines. This makes them a suitable choice for patients who are chronically hospitalized in intensive care units.

The benefits of midline catheters include a longer duration of use compared to peripheral catheters (up to 28 days), a lower incidence of procedure-related complications such as pneumothorax and infections and thrombosis compared to central lines. Moreover, they enable early removal of central lines and can be a viable option for patients with challenging vascular access, aiding in the preservation of venous reserve, which is often disregarded. These factors suggest that their use can result in decreased hospital costs. Unlike centrally inserted catheters, which require a physician's intervention for placement and removal, midline catheters can be inserted and removed by nursing professionals.

ELIGIBILITY:
Inclusion Criteria: Patients with prolonged hospitalization in ICU

-

Exclusion Criteria:

1. Pregnant women and terminal patients.
2. Skin infection at the site at the insertion site.
3. Central vascular occlusions, including patients with pacemakers.
4. Fistula for dialysis.
5. Mastectomy and lymphedema.
6. Positive blood cultures at the time of placement.
7. Coagulation disorders.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prolonged hospitalization in ICU (>10 days)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-03-20 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
infection reduction | 1 year
  Assessment of incidence of complications associated with midline catheters

SECONDARY OUTCOMES:
thrombosis reduction | 1 year
  Assessment of incidence of complications associated with midline catheters

CONTACTS AND LOCATIONS:
Overall Officials: Maximiliano Paz, BSN, Study Director — Hospital El Cruce
Locations (1):
- Hospital El Cruce, San Juan Bautista, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams DZ, Little A, Vinsant C, Khandelwal S. The Midline Catheter: A Clinical Review. J Emerg Med. 2016 Sep;51(3):252-8. doi: 10.1016/j.jemermed.2016.05.029. Epub 2016 Jul 5. PMID 27397766
- [Background] Zheng WM. Some exact results and approximations for cluster growth on the Cayley tree. Phys Rev A Gen Phys. 1987 Dec 15;36(12):5851-5853. doi: 10.1103/physreva.36.5851. No abstract available. PMID 9898877
- [Background] Hadaway L, Mermel LA. Midline Catheters: Could They Replace a Central Vascular Access Device? J Infus Nurs. 2022 Jul-Aug 01;45(4):220-224. doi: 10.1097/NAN.0000000000000471. PMID 35820127
- [Background] Terrault NA, Zhou S, Combs C, Hahn JA, Lake JR, Roberts JP, Ascher NL, Wright TL. Prophylaxis in liver transplant recipients using a fixed dosing schedule of hepatitis B immunoglobulin. Hepatology. 1996 Dec;24(6):1327-33. doi: 10.1002/hep.510240601. PMID 8938155